CLINICAL TRIAL: NCT02525822
Title: A Phase 2, Multi-Center, Double-Blind, Randomized, Vehicle-Controlled Study to Compare the Safety and Efficacy of IDP-123 Lotion to Tazorac® (Tazarotene) Cream, 0.1%, in the Treatment of Acne Vulgaris
Brief Title: Study to Compare the Safety and Efficacy of IDP-123 Lotion to Tazorac Cream in the Treatment of Acne Vulgaris
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Valeant Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V01-123A-201
Record Dates: First submitted 2015-08-13; First posted 2015-08-17 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — tazarotene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- IDP-123 Lotion (Experimental): IDP-123 Lotion, applied topically to the face, once daily for 12 weeks.
  Interventions: Drug: IDP-123 Lotion
- Tazorac Cream, 0.1% (Active Comparator): Tazorac Cream (tazarotene 0.1%), applied topically to the face, once daily for 12 weeks.
  Interventions: Drug: Tazorac Cream, 0.1%,
- Vehicle Cream (Placebo Comparator): Vehicle Cream, applied topically to the face, once daily for 12 weeks.
  Interventions: Drug: Vehicle Cream
- Vehicle Lotion (Placebo Comparator): Vehicle Lotion, applied topically to the face, once daily for 12 weeks.
  Interventions: Drug: Vehicle Lotion

INTERVENTIONS:
Drug: IDP-123 Lotion — Investigational Product: IDP-123 Lotion
  Arms: IDP-123 Lotion
Drug: Tazorac Cream, 0.1%, — Comparator Product: Tazorac Cream, 0.1%
  Other Names: tazarotene
  Arms: Tazorac Cream, 0.1%
Drug: Vehicle Cream — Comparator Product: Vehicle Cream
  Arms: Vehicle Cream
Drug: Vehicle Lotion — Comparator Product: Vehicle Lotion
  Arms: Vehicle Lotion

SUMMARY:
The primary objective of this study is to compare the safety and efficacy of once daily application of IDP-123 Lotion to Tazorac Cream, 0.1%, Vehicle Lotion, and Vehicle Cream in subjects with moderate to severe acne vulgaris.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, vehicle-controlled, 12-week study designed to assess the safety, tolerability, and efficacy of IDP-123 Lotion in comparison with Tazorac Cream, Vehicle Lotion, and Vehicle Cream in subjects with moderate to severe acne. Treatment success will be evaluated by changes in inflammatory and non-inflammatory lesion counts, as well as treatment success using an Evaluator's Global Severity Score. IDP-123 is a lotion for the topical treatment of acne.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 12 years of age and older
* Written and verbal informed consent must be obtained
* Subject must have a score of moderate or severe on the Evaluator's Global Severity assessment
* Pre-menses females and women of childbearing potential must have a negative urine pregnancy test at the screening and baseline visits
* Subjects must be willing to comply with study instructions and return to the clinic for required visits

Exclusion Criteria:

* Any dermatological conditions on the face that could interfere with clinical evaluations
* Any underlying disease(s) or some other dermatological condition of the face that requires the use of interfering topical or systemic therapy or makes evaluations and lesion count inconclusive
* Subjects with a facial beard or mustache that could interfere with the study assessments
* Subjects who are unable to communicate or cooperate with the Investigator
* Subjects with any underlying disease that the Investigator deems uncontrolled, and poses a concern for the subjects safety while participating in the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Absolute change in mean inflammatory lesion counts at Week 12 | 12 weeks
  Facial area lesion counts will be taken from the subject's face by the Evaluator at each visit and the change at week 12 from baseline will be calculated. Facial inflammatory lesions (pustules, papules, and nodules) will be counted as follows: pustules and papules will be counted and recorded together, not separately; nodular lesions will be counted and recorded separately.
  Inflammatory lesions are defined as follows:
  Papule - a solid, elevated lesion less than 5 mm; Pustule - an elevated lesion containing pus less than 5 mm; Nodule - palpable subcutaneous lesion greater than 5 mm; has depth, not necessarily elevated
Absolute change in mean non-inflammatory lesion counts at Week 12 | 12 weeks
  Facial area lesion counts will be taken from the subject's face by the Evaluator at each visit, and the change at week 12 from baseline will be calculated. Non-inflammatory lesions (open and closed comedones) will be counted and recorded together.
  Non-inflammatory lesions are defined as follows:
  Open comedones (blackhead) - plugged hair follicle with dilated/open orifice, black in color; Closed comedones (whitehead) - plugged hair follicle: small opening at skin surface
Percent of subjects who achieve at least a two-grade reduction from baseline and are Clear or Almost Clear at Week 12 in the Evaluator's Global Severity Score | 12 weeks
  At each visit the severity will be determined based on evaluator-blinded evaluations of the signs and symptoms of acne vulgaris. Evaluations will be scored on a scale of 0-4 (Evaluator's Global Severity Score), with 0 being clear and 4 being severe. Please see below for complete definitions.
  0 - Clear - Normal, clear skin with no evidence of acne vulgaris
  1. Almost clear- Rare non-inflammatory lesions present, with rare non-inflamed papules
  2. Mild- Some non-inflammatory lesions are present, with few inflammatory lesions (papules/pustules only; no nodulocystic lesions)
  3. Moderate-Non-inflammatory lesions predominate, with multiple inflammatory lesions evident: several to many comedones and papules/pustules, and there may or may not be one nodulocystic lesion
  4. Severe- Inflammatory lesions are more apparent, many comedones and papules/pustules, there may or may not be up to 2 nodulocystic lesions.

SECONDARY OUTCOMES:
Mean percent change in inflammatory lesion count from baseline at Weeks 2, 4, 8, and 12. | 2, 4, 8, and 12 weeks
  At each visit the Evaluator will count the total number of inflammatory lesions (papules, pustules, and nodules) on the subject's face, and the percent change will be calculated.
Mean percent change in non-inflammatory lesion counts from baseline at Weeks 2, 4, 8 and 12. | 2, 4, 8, and 12 weeks
  At each visit the Evaluator will count the total number of non-inflammatory lesions (open and closed comedones), and the percent change will be calculated.
The proportion of subjects with at least a two grade improvement in the Evaluator's Global Severity Score from baseline at Weeks 2, 4, 8 and 12. | 2, 4, 8, and 12 weeks
  At each visit the severity will be determined based on evaluator-blinded evaluations of the signs and symptoms of acne vulgaris. Evaluations will be scored on a scale of 0-4 (Evaluator's Global Severity Score), with 0 being clear and 4 being severe. Please see below for complete definitions.
  0 - Clear - Normal, clear skin with no evidence of acne vulgaris
  1. Almost clear- Rare non-inflammatory lesions present, with rare non-inflamed papules (papules must be resolving and may be hyperpigmented, though not pink-red)
  2. Mild- Some non-inflammatory lesions are present, with few inflammatory lesions (papules/pustules only; no nodulocystic lesions)
  3. Moderate-Non-inflammatory lesions predominate, with multiple inflammatory lesions evident: several to many comedones and papules/pustules, and there may or may not be one nodulocystic lesion
  4. Severe- Inflammatory lesions are more apparent, many comedones and papules/pustules, there may or may not be up to 2 nodulocystic lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, MS, Study Director — Valeant Pharmaceuticals